CLINICAL TRIAL: NCT04557124
Title: Understanding Social Situations (USS): Training to Improve Social Function in People With Psychosis
Brief Title: USS Training to Improve Social Function in People With Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3354-R
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Psychosis
Keywords: psychosis; social function; social cognition
MeSH Terms: conditions — Psychotic Disorders; Social Adjustment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- USS (Experimental): social cognitive training
  Interventions: Behavioral: USS
- MovingForward (Active Comparator): problem solving training
  Interventions: Behavioral: MovingForward

INTERVENTIONS:
Behavioral: USS — social cognitive training
  Arms: USS
Behavioral: MovingForward — problem solving training
  Arms: MovingForward

SUMMARY:
Psychotic spectrum disorders (PSD) are associated with poor social function. By doing this study, the investigators hope to learn which of two different types of 2-month long training courses is more effective in improving day-to-day interactions and quality of life.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of the two training courses. All participants will be asked to fill out questionnaires, engage in interviews, and complete paper and pencil tasks at the beginning of the study, at the halfway point of the training course (1 month), and end of the training course (2 months), and another 2 months later. One training focuses on how to make good judgments about what other people may be thinking or feeling in social situations, and why people might act in certain ways in different situations. The other training focuses on different strategies for handling everyday problems and stressors. Both trainings are done in one-on-one sessions with a research staff member. There will be 16-20 training sessions, each about 45-60 minutes long. The investigators will ask participants to attend 2 training sessions per week, so the total training time should be about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Veteran with diagnosis of psychotic disorder (e.g. schizophrenia, schizoaffective disorder, delusional disorder, psychosis NOS, etc);
* psychiatrically stable (30 or more days since last hospitalization/change in psychiatric medication)
* fluent in English
* able to provide legal written informed consent

Exclusion Criteria:

* current substance use disorder
* developmental disability
* severe, uncorrected auditory/visual impairment
* diagnosis of medical or neurological illness known to impair brain function including dementia, presence of seizures, history of head trauma with loss of consciousness > 1hr, or clear cognitive sequelae from other illness or injury
* currently enrolled in another treatment study targeting, or expected to impact, functioning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M. Fiszdon, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
see below
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available once primary and secondary study aims have been published.
Access Criteria: Completely de-identified data will be made available to other investigators, with written request and IRB approval, ideally under a data use agreement.

REFERENCES:
- [Derived] Fiszdon JM, Bell MD, Fulford D, Roberts DL, Dziura J, Parente L, Nasse A, Choi J. Understanding social situations: study protocol for a randomized controlled trial evaluating a novel social cognitive training versus modified problem-solving training for people with psychosis. Front Psychiatry. 2024 Aug 22;15:1440476. doi: 10.3389/fpsyt.2024.1440476. eCollection 2024. PMID 39238934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After obtaining consent but before randomization, 5 participants withdrew and 5 participants did not meet the inclusion criteria.
Groups:
- Understanding Social Situations (USS): social cognitive training
  USS: social cognitive training
- Moving Forward (MF): problem solving training
  MovingForward: problem solving training
Period: Allocation (Baseline)
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF)
Started | 53 | 50
Completed | 53 | 49
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Mid-point (1 Month)
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF)
Started | 53 | 49
Completed | 47 | 43
Not Completed | 6 | 6
Not completed — Missed testing | 5 | 4
Not completed — Lost to Follow-up | 1 | 2
Period: Post-testing (2 Months)
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF)
Started | 52 (Participants who missed testing appointments but did not lost to follow-up were allowed to participate in later testing.) | 47 (Participants who missed testing appointments but did not lost to follow-up were allowed to participate in later testing.)
Completed | 49 | 39
Not Completed | 3 | 8
Not completed — Missed testing | 1 | 5
Not completed — Lost to Follow-up | 2 | 3
Period: Follow-up (4 Months)
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF)
Started | 50 (Participants who missed testing appointments but did not lost to follow-up were allowed to participate in later testing.) | 44 (Participants who missed testing appointments but did not lost to follow-up were allowed to participate in later testing.)
Completed | 48 | 43
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Moving Forward (MF): Problem solving training
  Moving Forward: problem solving training
- Total: Total of all reporting groups
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF) | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [42 to 64] | 61 [47 to 68] | 60 [42 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 47 | 42 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 46 | 45 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 22 | 35
  White | 35 | 28 | 63
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Social Functioning Scale (SFS) [Median (Inter-Quartile Range); unit: units on a scale] — The SFS is one of the best known measures of social functioning in schizophrenia, and was one of two social function measures nominated by experts and selected by a RAND panel for a large-scale investigation of measures to assess real-world outcomes based on its psychometric properties, sensitivity to change, relationship to symptoms, and comprehensiveness. The total score ranges from 55 to 135, with a higher score indicates better social functioning.
  units on a scale | 105.57 [98.79 to 111.07] | 107.32 [99.50 to 111.57] | 105.79 [98.79 to 111.36]
Social Skill Performance Assessment (SSPA) [Median (Inter-Quartile Range); unit: units on a scale] — SSPA is a role-play measure of social skill ability. It consists of two, 3-minute, structured role plays (tenant meeting a new neighbor; tenant calling landlord to request repair). Each role play is rated between 1 and 5. The total score is calculated by summing up the ratings, and ranges from 2 to 10. A higher score indicates better social skill performance.
  units on a scale | 7.42 [7.13 to 8.40] | 7.38 [6.90 to 8.03] | 7.42 [7.01 to 8.25]

OUTCOME MEASURES:

1. Primary Outcome: Social Functioning Scale (SFS) Change
Description: The SFS is one of the best known measures of social functioning in schizophrenia, and was one of two social function measures nominated by experts and selected by a RAND panel for a large-scale investigation of measures to assess real-world outcomes based on its psychometric properties, sensitivity to change, relationship to symptoms, and comprehensiveness. The total score ranges from 55 to 135, with a higher score indicates better social functioning.
  Score change at post-testing (2 months) and follow-up (4 months) was calculated by subtracting the baseline score, with negative values indicating worse and positive values indicating better social functioning compared to baseline. Mid-testing (1 month) score change was included in the mixed-effects model, but its least square mean was not calculated as it was not a time point of interest.
Time Frame: Post-testing (2 months) and follow-up (4 months)
Population: An intention-to-treat analysis, including all randomized participants, was performed. A mixed-effects model was used to include all data points from randomization onward.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF)
Number analyzed (Participants) | 53 | 50
score on a scale
  Post-testing (2 months) | 1.28 [-0.04 to 2.59] | 0.19 [-1.22 to 1.60]
  Follow-up (4 months) | 1.56 [0.11 to 3.01] | 0.32 [-1.18 to 1.81]

2. Secondary Outcome: Social Skills Performance Assessment (SSPA) Change
Description: SSPA is a role-play measure of social skill ability. It consists of two, 3-minute, structured role plays (tenant meeting a new neighbor; tenant calling landlord to request repair). Each role play is rated between 1 and 5. The total score is calculated by summing up the ratings, and ranges from 2 to 10. A higher score indicates better social skill performance.
  Score change at post-testing (2 months) and follow-up (4 months) was calculated by subtracting the baseline score, with negative values indicating worse and positive values indicating better social skill performance compared to baseline.
Time Frame: Post-training (2 months) and follow-up (4 months).
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF)
Number analyzed (Participants) | 53 | 50
score on a scale
  Post-training (2 months) | 0.01 [-0.21 to 0.22] | -0.11 [-0.34 to 0.12]
  Follow-up (4 months) | 0.00 [-0.21 to 0.22] | -0.03 [-0.24 to 0.18]

ADVERSE EVENTS:
Time Frame: Up to 4 months.
Arm/Group | Understanding Social Situations (USS) | Moving Forward (MF)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 5/53 | 7/50
Other Adverse Events (participants affected / at risk) | 0/53 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Understanding Social Situations (USS) (N=53) | Moving Forward (MF) (N=50)
Heart failure exacerbation (Cardiac disorders) | 1 (1) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Delusions/Psychosis (Psychiatric disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Suicide ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Sprain and strain of ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Substance use (Psychiatric disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04557124/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04557124/ICF_000.pdf